CLINICAL TRIAL: NCT00183417
Title: Depression Prevention Program for High-Risk Adolescents
Brief Title: Depression Prevention Program for Adolescents
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas at Austin (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: R01MH067183 (NIH); R01MH067183 (NIH); DSIR 84-CTP
Record Dates: First submitted 2005-09-13; First posted 2005-09-16 (Estimated); Last update posted 2012-04-25 (Estimated); Status verified 2012-04

CONDITIONS: Depression
Keywords: Adolescent; CBT
MeSH Terms: conditions — Depression | interventions — Cognitive Behavioral Therapy; Palliative Care; Therapeutics; Bibliotherapy

ARMS (4):
- 1 (Experimental): Participants will receive cognitive behavioral therapy
  Interventions: Behavioral: Cognitive behavior therapy (CBT)
- 2 (Active Comparator): Participants will receive supportive/expressive therapy
  Interventions: Behavioral: Supportive/expressive (S/E) therapy
- 3 (Active Comparator): Participants will receive bibliotherapy
  Interventions: Behavioral: Bibliotherapy
- 4 (No Intervention): Participants in the control condition will receive no treatment

INTERVENTIONS:
Behavioral: Cognitive behavior therapy (CBT) — Participants will complete worksheets and group discussion on how to increase positive mood and activity.
  Arms: 1
Behavioral: Supportive/expressive (S/E) therapy — Participants will be encouraged to express feelings and emotions without advice giving.
  Arms: 2
Behavioral: Bibliotherapy — Participants will be given a book on how to increase their mood.
  Arms: 3

SUMMARY:
This study will compare the effectiveness of two programs designed to prevent depression in adolescents.

DETAILED DESCRIPTION:
Major depression is one of the most common psychiatric disorders in adolescents. In many cases, the condition is recurrent and can result in serious psychological impairment. A high number of depressed adolescents never receive treatment; therefore, it is crucial to develop prevention programs for this disorder that are effective and can be easily disseminated. This study will evaluate and compare the effectiveness of cognitive behavior therapy (CBT) and supportive/expressive (S/E) therapy in preventing depressive symptoms in adolescents.

This study will last 2 years. Participants will be randomly assigned to receive six sessions of CBT, S/E therapy, or standard depression education over 2 years. The CBT intervention will focus on reducing negative thoughts and increasing engagement in pleasant activities. S/E therapy is designed to allow adolescents to express their negative emotions and talk about recent stressful events in a supportive environment of their peers. Surveys and psychiatric interviews will be completed by all participants and their parents at the beginning and the end of the study. The surveys and interviews will assess depressive symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Beck Depression Inventory score higher than 10
* Parent or guardian willing to provide informed consent

Exclusion Criteria:

* Diagnosis of depression

Ages: 14 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 350 (Actual)
Dates: Start 2004-09; Primary Completion 2009-05 (Actual); Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
Depressive symptoms | Measured at Year 1

CONTACTS AND LOCATIONS:
Overall Officials: Eric M. Stice, PhD, Principal Investigator — University of Texas at Austin
Locations (1):
- University of Texas at Austin, Austin, Texas, United States

REFERENCES:
- [Derived] Gau JM, Stice E, Rohde P, Seeley JR. Negative life events and substance use moderate cognitive behavioral adolescent depression prevention intervention. Cogn Behav Ther. 2012;41(3):241-50. doi: 10.1080/16506073.2011.649781. Epub 2012 Mar 13. PMID 22414236